CLINICAL TRIAL: NCT06060522
Title: Multi-detector Computed Tomography Versus Cone Beam Computed Tomography as a Diagnostic Imaging in Retrieval of Displaced Mandibular Third Molar Teeth/Roots
Brief Title: Retrieval of Displaced Mandibular Third Molar Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Kamal Eid Allam, Associate professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M22011122
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Tooth Displacement
Keywords: Displaced wisdom; Computed Tomography; Cone beam Computed Tomography

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-detector computed tomography (MDCT ) (Active Comparator): Multi-detector computed tomography (MDCT ) will be performed for 8 patients performed using CT scanner (SOMATOM Emotion6, Siemens, Germany). The protocol was 200 mAs, 120 kVp, 512 × 512 matrix, 1.172 pitch, 64 × 0.625 mm section collimation, 2 mm slice thickness, 0.6 mm section reconstruction
  Interventions: Diagnostic Test: CT, CBCT
- CBCT scans (Active Comparator): CBCT will be performed for 8 patients with an exposure performed at 15 mA, 85 KV and at a field of view 7.5 cm x 14.5 cm x 14.5 cm.
  Interventions: Diagnostic Test: CT, CBCT

INTERVENTIONS:
Diagnostic Test: CT, CBCT — Under general anesthesia, a lingual envelope incision is performed to access and remove the displaced third molar tooth or root, and a mucoperiosteal flap is released from the retromolar trigone to the medial surface of the mandibular first premolar. By carefully retracting the lingual soft tissue, an envelope flap is raised on the lingual side from the second premolar to the anterior boundary of the ramus. This protected the lingual nerve from injury. With great caution, the lingual flap is reflected up to the submandibular area so that the tooth or root fragment will be identified. An extra-oral finger is used as support.Through blunt dissection, the loose tooth or root is located, grabbed using a pair of artery forceps, and extracted.
  The flaps are sutured using 3-0 Vicryl sutures after the wound is irrigated with normal saline.
  Other Names: Surgery

SUMMARY:
The aim of this study is to compare multi-detector CT and CBCT as pre-surgical diagnostic imaging before surgical retrieval of iatrogenic displaced mandibular third molar teeth/roots.

DETAILED DESCRIPTION:
Sixteen patients will included in this study that they had previously a challenging and unsuccessful extraction of an impacted mandibular third molar by a general dentist under local anesthesia.

Groups allocation:

For detailed radiographic examination, when a displaced tooth/root fragment is suspected the patients will randomly divided into two equal groups, each of eight patients:

Group (1): Multi-detector computed tomography (MDCT ) are performed using CT scanner (SOMATOM Emotion6, Siemens, Germany). The protocol is 200 mAs, 120 kVp, 512 × 512 matrix, 1.172 pitch, 64 × 0.625 mm section collimation, 2 mm slice thickness, 0.6 mm section reconstruction Group (II): CBCT** scans are performed with an exposure performed at 15 mA, 85 KV and at a field of view 7.5 cm x 14.5 cm x 14.5 cm.

Image reconstruction All images will be reconstructed at 0.6 mm and the reconstructed axial images are transferred to a workstation, and multi-planar reconstructions are generated using the included standard dental software package. The panoramic and paraxial images were obtained perpendicular to the transverse images. Then multi-planar reformation (MPR), maximum intensity projection (MIP) and shaded surface display (SSD) are done in different planes.

Image interpretation (analysis):

Axial and reformatted images are evaluated to detected the position of displaced third molar tooth or root in relation to the mandible and the mylohyoid muscle.

Preoperative instruction It will intended for all patients to have their displaced tooth or root fragments retrieved using an intra-oral approach while being under general anesthesia following standard blood tests and pre-anesthetic examinations.

Surgical procedure All surgeries are performed in a standardized fashion, using the same surgical and pharmacological protocols. All surgeons had at least 5 years of experience in third molar teeth extraction. Before surgery, the patient performed a mouth rinse of chlorhexidine 0.12% for one minute. Dexamethasone 8 mg is given orally to the patient one hour before surgery to promote the best possible postoperative results.

Under general anesthesia, a lingual envelope incision is performed to access and remove the displaced third molar tooth or root, and a mucoperiosteal flap was released from the retromolar trigone to the medial surface of the mandibular first premolar. By carefully retracting the lingual soft tissue, an envelope flap was raised on the lingual side from the second premolar to the anterior boundary of the ramus. This protected the lingual nerve from injury. With great caution, the lingual flap is reflected up to the submandibular area so that the tooth or root fragment will be identified. An extra-oral finger is used as support. (Jo Through blunt dissection, the loose tooth or root is located, grabbed using a pair of artery forceps, and extracted. The flaps are sutured using 3-0 Vicryl sutures after the wound was irrigated with normal saline.

Post-operative evaluation At the conclusion of the intervention, the same operators meticulously filled out a data collection form for each patient. These documents are momentarily kept in a secure location inside the operational unit. A progressive numerical code is given to each patient as a means of identification. Gender, birthdate, the anatomical location of the misplaced tooth or root, and the duration of the operation (calculated from the incision to socket cleaning) are all collected.

On the seventh post-operative day, the sutures are removed, and the patients are evaluated for the following: Pain , swelling ,Trismus and Sensory disturbances

ELIGIBILITY:
Inclusion Criteria:

- Patients had a challenging and unsuccessful extraction of an impacted mandibular third molar by a general dentist under local anesthesia.

Exclusion Criteria:

* Patients presented with pathologic lesions (dental cyst or tumor) around the tooth to be retrieved

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
degree of Pain | 3 months
  The degree of pain is determined during the follow-up periods according to the visual analogue pain scale (VAS) from 0 (no pain at all) to 10 (most severe pain)
Swelling | 3 months
  assessed utilizing a vertical and horizontal guide with a tape on four reference points; outer canthus of the eye, angle of the mandible, tragus, and outer corner of the mouth respectively
Sensory disturbances | 3 months
  Nerve dysesthesia is recorded using two-point discrimination test

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed K Allam, Ass prof, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No